CLINICAL TRIAL: NCT06686472
Title: A Single-Center, Randomized, Double-masked, Vehicle-controlled Phase 2 Study Evaluating the Safety and Efficacy of TL-925 Ophthalmic Emulsion 0.1% Compared to Vehicle for the Treatment of Allergic Conjunctivitis in the Conjunctival Allergen Challenge (Ora-CAC®) Model
Brief Title: Evaluation of TL-925 for the Treatment of Allergic Conjunctivitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TL-925-308
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sponsor, investigators, and study staff will be masked throughout the study. The study site will have the capacity to unmask in case of emergency. Following completion of the study, the randomization code will be unmasked once all data has been entered into the study database for every subject, and the database has been locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TL-925 Arm (Active Comparator): Subjects will be dosed in clinic.
  Interventions: Drug: TL-925
- Placebo Arm (Placebo Comparator): Subjects will be dosed in clinic.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TL-925 — TL-925 is an eye drop.
  Arms: TL-925 Arm
Drug: Placebo — The composition of the placebo is identical to the active formulation except for the exclusion of the active ingredient.
  Arms: Placebo Arm

SUMMARY:
In this prospective, Phase 2, randomized, double-masked, vehicle controlled study, approximately 66 eligible subjects will be randomized 1:1 to receive either TL-925 or placebo as topical ophthalmic eye drops administered bilaterally.

The study comprises of a screening and treatment period using the conjunctival allergen challenge model to evaluate TL-925 for the treatment of allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* Female subjects of childbearing potential and their male partners must both use a highly effective contraception method during the study.
* Documented history of ocular allergies and a positive skin test reaction to a seasonal (grass, ragweed, tree pollen) or perennial (cat dander, dog dander, dust mites, cockroach) allergen as confirmed by an allergic skin test conducted at Visit 1 or within the past 60 months.
* Calculated best-corrected visual activity of 0.7 LogMAR or better
* Positive bilateral CAC reaction

Exclusion Criteria:

* Any systemic or ocular disease currently producing ocular redness and/or ocular discomfort, or that may interfere with the conduct of the study.
* Any ocular surgical intervention within the last 3 months OR refractive surgery within the last 6 months
* Any ongoing ocular infection (bacterial, viral or fungal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Ocular Itching | 3, 5 and 7 minutes after CAC
  Ocular itching score will be reported by the subject at 3 timepoints after CAC at Visits 4b , 5, and 6b. Assessments are reported using a 0-4 numerical scale (0 = none and 4 = incapacitating itch with an irresistible urge to rub).
Conjunctival Redness | 7, 15 and 20 minutes after CAC
  Conjunctival redness score will be evaluated by the investigator at 3 timepoints after CAC at Visits 4b, 5, and 6b. Assessments are completed using a 0-4 numerical scale (0 = none and 4 = extremely severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Telios Investigative Site, Memphis, Tennessee, United States